CLINICAL TRIAL: NCT07398391
Title: Blood Pressure Care for Advancing Real-World Evidence (BPCARE): an RCT of Adherence
Brief Title: Blood Pressure Care for Advancing Real-World Evidence (BPCARE)
Acronym: BPCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Family Health Centers of San Diego (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tala A lRousan, Assistant Adjunct Professor, Herbert Wertheim School of Public Health & Human Longevity Science, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHRC-BPCARE; 1R01HL173155-01A1 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; High Blood Pressure
Keywords: Medication Adherence; Chronic Disease Management; Blood Pressure Self-Management; Federally Qualified Health Center; Motivational Interviewing
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPCARE Intervention Arm (Experimental): Participants in the BPCARE intervention arm will receive a translated educational booklet, a pill box for pill organization, and two intervention sessions focused on medication adherence within month 1 and 2 after randomization.
  Interventions: Behavioral: BPCARE Intervention
- Standard Care Control Arm (No Intervention): Participants in the control arm will not receive any additional support, but will still be conducting monthly pill counts, at home BP measurements, and in-person follow-up visits.

INTERVENTIONS:
Behavioral: BPCARE Intervention — Participants randomized to the BPCARE intervention will receive a culturally and linguistically tailored hypertension-education booklet, a pill organizer to support medication adherence, and two structured intervention sessions focused on medication adherence delivered within month 1 and 2 after randomization. These sessions include individualized counseling on blood pressure management, medication adherence strategies, and lifestyle modification. Participants will also receive ongoing follow-up and support from trained Patient Health Navigators (PHNs), including check-ins, problem-solving assistance, and linkage to additional resources as needed.
  Other Names: BPCARE
  Arms: BPCARE Intervention Arm

SUMMARY:
The goal of this randomized clinical trial is to determine whether a community health worker-delivered, multi-component behavioral intervention can improve antihypertensive medication adherence and blood pressure control among adult refugees with hypertension who are prescribed antihypertensive medications.

The main questions it aims to answer are:

1. Does participation in the BPCARE intervention improve antihypertensive medication adherence compared to enhanced usual care?
2. Does participation in the BPCARE intervention improve blood pressure control and persistence over time compared to enhanced usual care?

Researchers will compare participants randomized to the BPCARE intervention to those receiving enhanced usual care (hypertension information and a home blood pressure monitor) to determine the effects on medication adherence, blood pressure control, and persistence.

Participants will:

* Be randomly assigned to either the BPCARE intervention or enhanced usual care
* Receive hypertension education and a home blood pressure monitor
* Participate in community health worker-delivered sessions that include hypertension and medication education, motivational interviewing, problem-solving, and action planning (intervention arm only)
* Complete questionnaires assessing medication adherence and related psychosocial factors
* Have blood pressure monitored using connected home blood pressure devices
* Complete pill counts to assess medication adherence over a nine-month follow-up period

DETAILED DESCRIPTION:
Blood Pressure Care for Advancing Real-World Evidence (BPCARE) is a randomized controlled study conducted within a federally qualified health center (FQHC) to examine a community health worker-delivered behavioral intervention integrated into routine hypertension care. The study is implemented at Family Health Centers of San Diego (FHCSD), a safety-net healthcare system serving patients with diagnosed hypertension.

Uncontrolled blood pressure remains a major contributor to cardiovascular morbidity, particularly among patients who experience challenges such as language discordance, limited resources, and healthcare access difficulties. Team-based care approaches that extend beyond physician-led models are increasingly used in clinical practice to support hypertension management. Non-physician-led behavioral strategies, including interventions delivered by community health workers (CHWs), have demonstrated potential to support medication-taking behaviors by facilitating patient engagement and connection with the healthcare system.

Participants complete screening and baseline assessments prior to randomization. Following randomization, participants are considered enrolled and are followed for a total of six months. A total of 250 patients with a diagnosis of hypertension receiving care at FHCSD will be assigned in a 1:1 ratio to either the BPCARE intervention or standard medical care. Study activities include a pre-randomization orientation/baseline visit, in-person follow-up visits at three and six months, and monthly unannounced pill count video visits.

During the pre-randomization orientation/baseline visit, participants receive a detailed overview of study procedures, provide informed consent, complete baseline questionnaires, undergo an initial pill count, and receive training on conducting monthly pill counts and measuring blood pressure at home using study-provided devices.

Participants assigned to the intervention arm receive structured support from trained community health workers during the first three months of study participation. Community health workers deliver culturally tailored, theory-informed educational and behavioral strategies, including hypertension and medication education, motivational interviewing, problem-solving and action planning, and ongoing medication adherence support.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of hypertension determined at screening,
* Be at least 21 years of age,
* English as a second language,
* Be able to provide written informed consent and participate in study procedures,
* Have a last least one recorded automated clinic systolic BP reading of at least 130 mmHg within the past year OR at least one home SBP reading of ≥140 mmHg in the last year. AND/OR answer is in range of less than two months to "when was the last time you missed a dose of your hypertension medication?"
* Will not move out of San Diego in the next 6 months, and
* Have access to a mobile phone or computer with video telecommunication capacity (e.g. Zoom)

Exclusion Criteria:

* A cardiovascular event or hospitalization for unstable angina within last 3 months,
* Symptomatic heart failure within the past 6 months or left ventricular ejection fraction < 35%,
* Individuals who are pregnant, planning on becoming pregnant within the next 7 months
* Current participation in another clinical trial that includes taking medications that may change blood pressure, or
* Major factors judged to be likely to significantly limit comprehension of or adherence to interventions including dementia, psychotic disorders, or affect ability to conduct pill counts
* Any immediate family members participating in the trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Assessed by Self-Report Questionnaire and Unannounced Pill Counts | From baseline/orientation until the end of the follow-up visit at 6 months post randomization
  Test the efficacy of BPCARE in improving antihypertensive medication adherence at 6 months post randomization (primary outcome; via self-report (Hill-Bone Compliance questionnaire), and unannounced pill counts (using video telecommunications)) compared to enhanced usual care. Hypotheses: BPCARE improves antihypertensive medication adherence H1a through H1b increased hypertension and medication adherence knowledge, H1c increased disease risk perceptions and therapeutic interest and motivation, H1d increased self-efficacy and behavioral skills, H1e reduced barriers, H1f long-term persistence (i.e., time to medication self-discontinuation at 6 months post randomization).

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure Measured by Connected Blood Pressure Cuff | From baseline/orientation until the end of the follow-up visit at 6 months post randomization
  Test the efficacy of BPCARE in improving systolic blood pressure at 6 months post randomization (secondary outcome via connected BP cuffs) among hypertensive refugees compared to enhanced usual care. H2: More refugees will have controlled BP in the BPCARE group compared to the control group at 6 months post randomization.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Family Health Centers of San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No